CLINICAL TRIAL: NCT03566914
Title: A Randomized Placebo Controlled Trial of Tadalafil for Erectile Dysfunction in Patients With Cirrhosis
Brief Title: Tadalafil for Erectile Dysfunction in Patients With Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-16
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tadalafil (Experimental): Tadalafil 10 mg once daily per oral for 3 months
  Interventions: Drug: Tadalafil 10 MG
- Placebo (Placebo Comparator): Tablet placebo once daily per oral for 3 months
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tadalafil 10 MG — Tadalafil 10 mg per oral once daily for 3 months
  Arms: Tadalafil
Other: Placebo — TPlacebo tablet per oral once daily for 3 months
  Arms: Placebo

SUMMARY:
This study will be conducted into two parts 1) Screening of 400 cases of cirrhosis (Child A,child B and child c) for the prevalence and risk factors of erectile dysfunction in cirrhosis.2) The part 2 is RCT as follows where 70 cases in each arm will be taken wuth child A and child B cirrhosis for the effect of treatment on erectile dysfunction (Tadalafil vs Placebo).

After getting informed consent. Clinical, anthropometric and biochemical assessment will be done by candidate, co-supervisors and supervisor. Screening and selection criteria by using various questionnaire like Karnofsky Performance Score (KPS) , IIEF Questionnaire , ADAMS Questionnaire, Generalized Anxiety Disorder 7 (GAD-7) questionnaire, Patient Health Questionnaire (PHQ-9 for depression ; and SF-36 questionnaire).

The informed consent will be obtained from the participants in the study. Patients-ED IIEF<25 will be included as per inclusion and exclusion criteria. Tadalfil regimen: 10 mg daily at any time before anticipated sexual activity on days with anticipated sexual activity On days with no anticipated sexual activity: 10 mg daily at night after meals. Follow-up1 week, 2weeks, 4weeks, 12 weeks with history, clinical examination and laboratory test.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients, age from 21 years to 60 years ;
2. Child´s Grade A or B cirrhosis (CTP score up to 9) of any etiology;
3. A minimum 3-month history of mild-to-severe ED;
4. A stable monogamous relationship with a female partner and anticipate having same adult female sexual partner during the study.
5. Sexually active- They should also agree to make at least 4 sexual intercourse attempts with the female partner during the 4-week run-in phase without medication; agree to make at least 1 sexual intercourse attempt per day with the female partner during days 1-4 following randomization (with a minimum of three attempts required during that period). Also agree to make at least 3 intercourse attempts during days 5-14 following randomization.
6. Men with a history of hypertension, hypercholesterolemia and diabetes will be included.
7. Following beta-blocker therapy was allowed: Carvedilol (up to the max. dose of 25 mg) and propranolol (up to the max. dose of 160 mg).
8. Patients will be included if they were not on beta-blocker or on a stable dose of beta-blocker for at least last 6 weeks ( beta-blocker dose was not modified during the duration of the study).
9. Patients with history of endoscopically diagnosed large esophageal varices without previous bleeding will be included if they were on a stable dose of prophylactic beta blocker for at least last 6 weeks ( beta-blocker dose was not modified during the duration of the study) or on endoscopic band ligation sessions ( should have small esophageal varices at the time on enrollment in the study, and the last endoscopic band ligation session at least >1 week ago).

Exclusion Criteria:

1. Patients with overt hepatic encephalopathy; Child´s grade C cirrhosis; history of variceal bleeding within last 4 weeks [ patients were included if they bled >4 weeks ago and were on secondary prophylaxis with endoscopic band ligation( should have small esophageal varices at the time on enrollment in the study, and the last endoscopic band ligation session at least >1 week ago) and/or beta-blockers ; and hepatocellular carcinoma; acute decompensated state of cirrhosis like gastrointestinal bleed/increased jaundice, active infection, post TIPS patients, acute febrile illness excluded.
2. Patients with HbA1c >13.0% at the screening visit (visit 1, week -4), a recent history of diabetic ketoacidosis (≥ 2 episodes), or ≥ 3 episodes of hypoglycemia requiring assistance were excluded. However, men with microvascular complications, including retinopathy, were eligible.
3. Patients with history of angina during intercourse, unstable angina, or any other evidence of recently diagnosed coronary artery disease, poorly controlled blood pressure (systolic >170 or_<90mm Hg or diastolic _>100 or _<50 mmHg) or orthostatic hypotension, arrhythmia, uncontrolled congestive heart failure, renal or respiratory failure, and anemia were also excluded.
4. Men who failed to achieve an erection after radical prostatectomy or pelvic surgery; those who had penile implants, clinically noteworthy penile deformities, or a history of psychiatric disorders, stroke or spinal-cord trauma within 6 months of study onset; those who were receiving nitrates, antiandrogens, antidepressant, anticonvulsants, other hypnotics or cancer chemotherapy; and patients with active alcohol intake or intake within 1 month of enrollment, active substance abuse or intake within 1 month of enrollment also excluded.
5. Patients with history of hypersensitivity to the trial drugs or to drugs with a similar chemical structure,
6. Patients with Karnofsky performance status of below 70% were excluded
7. Patient with uncontrolled thyroid disorders.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2019-12-28 (Actual)

PRIMARY OUTCOMES:
Proportions of patients achieving more than a five-point gain from baseline to end point in the erectile function domain of the IIEF ( International Index of Erectile Function). | 3 Months

SECONDARY OUTCOMES:
Number of patients with erectile Dysfunction | 1.5 years
Side effects of tadalafil drug | 3 months
Reduction in HVPG (Hepatic Venous Pressure Gradient) ≥10 in both groups | 3 Months
Change in Sexual Encounter Profile (SEP) in both groups | 3 Months
Global Assessment Index in both groups | 3 Months
Improvement in q ADAMS in both groups | 3 Months
Improvement in PHQ 9 in both groups | 3 Months
Improvement in GAD 7 in both groups | 3 Months
Improvement in SF-36 in both groups | 3 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Rakesh Kumar Jagdish, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jagdish RK, Kamaal A, Shasthry SM, Benjamin J, Maiwall R, Jindal A, Choudhary A, Rajan V, Arora V, Bhardwaj A, Kumar G, Kumar M, Sarin SK. Tadalafil improves erectile dysfunction and quality of life in men with cirrhosis: a randomized double blind placebo controlled trial. Hepatol Int. 2023 Apr;17(2):434-451. doi: 10.1007/s12072-021-10264-w. Epub 2021 Nov 14. PMID 34775577